CLINICAL TRIAL: NCT05912010
Title: A Study on Pathogenic Surveillance and Nasopharyngeal Carriage of Children and Adolescents Based on Hospitals and Communities in Hainan Province
Status: Completed | Type: Observational
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Director of Division of Infectious Diseases Affiliation: Huashan Hospital, Huashan Hospital
Other Study IDs: HAPEC-Stage one 01&02
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2023-06

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- case group: patients from fever clinics and pediatric wards
  Interventions: Diagnostic Test: NP/OP swab
- control group: healthy community children
  Interventions: Diagnostic Test: NP/OP swab

INTERVENTIONS:
Diagnostic Test: NP/OP swab — NP/OP (nasopharyngeal/oropharyngeal) swabs will be collected from all cases at enrollment for respiratory pathogen multiplex PCR or pneumococcus culture.

SUMMARY:
This study intends to screen children under the age of 10 for respiratory pathogens, Streptococcus pneumoniae, and serotyping in three representative cities in Hainan province: Haikou, Wanning, and Baisha, in order to provide a foundation for the subsequent promotion of Streptococcus pneumoniae vaccines.

DETAILED DESCRIPTION:
The purpose of this multi-center epidemiological study was to determine the carrier status of clinically diagnosed pneumonia, pathogen spectrum of clinically diagnosed pneumonia, serotype distribution, and drug resistance profile of Streptococcus pneumoniae in sick children from hospitals and healthy children from the community.

ELIGIBILITY:
Inclusion Criteria:

* 1. Case group: patients from fever clinics and pediatric wards

Patients with at least one of the following will be clinically diagnosed with pneumonia and recommended for NP/OP, blood cultures, or induced sputum as clinically indicated (TB only or if performed routinely by the clinician), bronchoalveolar lavage fluid (BALF , according to clinical requirements), pleural effusion (according to clinical requirements), and chest X-ray examination:

1. Shortness of breath ( children <2 months, respiratory rate ≥60 breaths/min; children ≥2 months to <12 months, respiratory rate ≥50 breaths/min; children ≥12 months to < 60 months, respiratory rate ≥40 breaths/min; Children ≥ 60 months to < 120 months, respiratory rate > 24 breaths/minute )
2. Rales on lung auscultation
3. Respiratory symptoms and fever ( axillary temperature ≥ 37.5 ℃ or rectal temperature ≥ 38 ℃ )

   * 2. Control group The control group will be randomly selected from the community and frequency-matched 1:1 with the case group according to age group, sex and city.

Exclusion Criteria:

* 1. Hospitalized within the first 14 days, or discharged as a case group within the first 30 days, and lived outside the research center area ;
* 2. People who affect the research results: patients cannot keep samples or the amount of samples is not enough for testing;
* 3. Can't cooperate well;
* 4. The researcher judges that it is not suitable to be included in this study .

Ages: 1 Month to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The prevalance of clinial diagnosed pneumonia and invasive diseases in Hainan Province will be mainly collected from the electronic medical record (EMR) database of selected hospitals and face-to-face questionnaire survey, in the fever clinics and pediatric wards of selected hospitals. A control group of healthy community children will be systematically sampled from residents from the same area as the cases and frequency-matched by age group.
Sampling Method: Probability Sample
Enrollment: 3746 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of pneumococcus | 1 day
  Estimate the prevalence of pneumococcus among children aged<10 years old hospitalized with clinical diagnosed pneumonia, in children seen at outpatient clinics, and among healthy children in the community in Hainan
Correaltion index of high load (>6.9 log10 copies/ml) pneumococcus | 1 day
  Estimate the association with disease (i.e., case-control status) of high load (>6.9 log10 copies/ml) pneumococcus among outpatient or hospitalized patients with clinical diagnosed pneumonia in children aged<10 years old and among healthy children in the community in Hainan
Correaltion index of disease status of infection with different pathogens | 1 day
  Estimate the association with disease status of infection with pathogens of interest (or combination of pathogens) among children aged<10 years old hospitalized with clinical diagnosed pneumonia compared to healthy children in the community in Hainan. The study is designed to be the case-control study

SECONDARY OUTCOMES:
Estimate the proportions of srotypes in patients and healthy children | 1 day
  Estimate the pneumococcal serotype distribution in children aged<10 years old with clinically diagnosed pneumonia carrying pneumococcus in Hainan.
Describe the resistance proportion of antibiotics in different region in Hainan | 1 day
  Describe the antimicrobial resistance patterns in children aged<10 years old with clinically diagnosed pneumonia carrying pneumococcus in Hainan.

CONTACTS AND LOCATIONS:
Overall Officials: Wenhong Zhang, M.D., Principal Investigator — Huashan Hospital
Locations (5):
- China (5):
  - People's Hospital of Baisha Li Autonomous County, Baisha, Hainan
  - Haikou Hospital of the Maternal and Child Health, Haikou, Hainan
  - Hainan Women and Childrens Medical Center, Haikou, Hainan
  - The First Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - People's Hospital of Wanning, Wanning, Hainan

IPD SHARING:
Plan to Share IPD: Undecided
After thesis defense the study may be published internationally to be available for the public.

REFERENCES:
- [Background] Alizadeh Chamkhaleh M, Esteghamati A, Sayyahfar S, Gandomi-Mohammadabadi A, Balasi J, Abdiaei H, Moradi Y, Moradi-Lakeh M. Serotype distribution of Streptococcus pneumoniae among healthy carriers and clinical patients: a systematic review from Iran. Eur J Clin Microbiol Infect Dis. 2020 Dec;39(12):2257-2267. doi: 10.1007/s10096-020-03963-z. Epub 2020 Jun 29. PMID 32601893
- [Background] Hocknell RE, Cleary DW, Srifeungfung S, Clarke SC. Serotype distribution of disease-causing Streptococcus pneumoniae in Thailand: A systematic review. Vaccine. 2019 May 27;37(24):3159-3166. doi: 10.1016/j.vaccine.2019.04.085. Epub 2019 May 3. PMID 31060951
- [Background] Jauneikaite E, Jefferies JM, Hibberd ML, Clarke SC. Prevalence of Streptococcus pneumoniae serotypes causing invasive and non-invasive disease in South East Asia: a review. Vaccine. 2012 May 21;30(24):3503-14. doi: 10.1016/j.vaccine.2012.03.066. Epub 2012 Apr 1. PMID 22475858
- [Background] Andrejko K, Ratnasiri B, Hausdorff WP, Laxminarayan R, Lewnard JA. Antimicrobial resistance in paediatric Streptococcus pneumoniae isolates amid global implementation of pneumococcal conjugate vaccines: a systematic review and meta-regression analysis. Lancet Microbe. 2021 Sep;2(9):e450-e460. doi: 10.1016/S2666-5247(21)00064-1. PMID 34485957
- [Background] Lyu S, Hu HL, Yang YH, Yao KH. A systematic review about Streptococcus Pneumoniae serotype distribution in children in mainland of China before the PCV13 was licensed. Expert Rev Vaccines. 2017 Oct;16(10):997-1006. doi: 10.1080/14760584.2017.1360771. Epub 2017 Aug 9. PMID 28745918
- [Background] Zhao C, Zhang F, Chu Y, Liu Y, Cao B, Chen M, Yu Y, Liao K, Zhang L, Sun Z, Hu B, Lei J, Hu Z, Zhang X, Wang H. Phenotypic and genotypic characteristic of invasive pneumococcal isolates from both children and adult patients from a multicenter surveillance in China 2005-2011. PLoS One. 2013 Dec 11;8(12):e82361. doi: 10.1371/journal.pone.0082361. eCollection 2013. PMID 24349263
- [Background] DeVries A, McCauley K, Fadrosh D, Fujimura KE, Stern DA, Lynch SV, Vercelli D. Maternal prenatal immunity, neonatal trained immunity, and early airway microbiota shape childhood asthma development. Allergy. 2022 Dec;77(12):3617-3628. doi: 10.1111/all.15442. Epub 2022 Jul 25. PMID 35841380